CLINICAL TRIAL: NCT05249608
Title: A Prospective, Open-label, Multicenter, Single-arm Clinical Study to Evaluate the Safety and Performance of the Gastric Bypass Stent System as a Weight Loss Treatment for Obesity
Brief Title: Tangji EU Gastric Bypass Stent Study for Obesity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hangzhou Tangji Medical Technology Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BL-RD08-040
Record Dates: First submitted 2022-01-18; First posted 2022-02-21 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Adiposity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Other): A single arm study, only investigational product-the Gastric Bypass Stent System is intended to be used in weight loss treatment for obesity in patients with a BMI ≥ 30 kg/m2. to evaluate the safety and performance of the investigational device for the intended use.
  Interventions: Device: A prospective, open-label, multicenter, single-arm clinical study to evaluate the safety and performance of the Gastric Bypass Stent System as a weight loss treatment for obesity

INTERVENTIONS:
Device: A prospective, open-label, multicenter, single-arm clinical study to evaluate the safety and performance of the Gastric Bypass Stent System as a weight loss treatment for obesity — This study includes 3 phases; screening period, procedural period, and a follow-up period. Following a 2-week screening period, subjects will be treated with the Gastric Bypass Stent System implanted under gastroscopy (Visit 2; Day 0). Following a 3-month treatment period, the device is removed, and subjects are followed for 6 months. In total subject participation will last for approximately 9 months.

SUMMARY:
The Gastric Bypass Stent System is intended to be used in weight loss treatment for obesity in patients with a BMI ≥ 30 kg/m2. In this clinical investigation the Sponsor seeks to demonstrate the safety and performance of the Gastric Bypass Stent System for its proposed indication in weight loss treatment for obesity in the European Union (EU) and United Kingdom (UK).

DETAILED DESCRIPTION:
The Gastric Bypass Stent System is intended to be used in weight loss treatment for obesity in patients with a BMI ≥ 30 kg/m2. In this pivotal, prospective, multicenter, single-arm clinical investigation the Sponsor seeks to demonstrate the safety and performance of the Gastric Bypass Stent System for its proposed indication in weight loss treatment for obesity in the European Union (EU) and United Kingdom (UK). This clinical investigation will be used as an EU/UK bridging study and, with the ongoing clinical investigation in China (Protocol number: HZTG01), will be used to evaluate the safety and performance of the investigational device for the intended use.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female aged 18 to 60 years old.
* Obese patients with BMI ≥ 30 kg/m2, who are willing to be treated with Gastric Bypass Stent System.
* Patients with American Society of Anesthesiologists (ASA) I~II grade. Exception: patients with BMI ≥ 40 kg/m2 may be included upon the Investigator's discretion if they have no other severe systemic disease.
* Able and willing to provide informed consent for participation in the clinical investigation and comply with all study procedures and assessments.

Exclusion Criteria:

* Have lost more than 4.5 kg in the past three months or have taken weight loss drugs in the past month.
* Patients with secondary obesity; a medical condition that has caused weight gain such as endocrine disorders and hypothalamic disorders.
* Chronic, daily use of systemic anti-inflammatory or corticosteroid medications (e.g., ibuprofen, prednisolone) for more than 1 week (not including low-dose aspirin for cardiac prophylaxis or inhaled corticosteroids).
* Patients with less than one-year continuous treatment before baseline with hypoglycemic drugs with known weight loss effects (e.g., GLP-1 agonists, SGLT-2 inhibitors, DDP-4 inhibitors).
* Patients diagnosed with type 1 diabetes.
* Patients with the function of islet β cell basically lost, C-peptide ≤ 1/2 of the normal low limit, or low and flat C-peptide release curve under glucose load.
* Patients with significant iron deficiency or iron deficiency anemia upon the Investigator's discretion.
* Patients with coagulation dysfunction and chronic, daily use of systemic anti-inflammatory or anti-coagulation medication in the past month (not including low-dose aspirin).
* Patients with severe liver and kidney dysfunction, and a serum creatinine concentration ≥ 180 μmol/L.
* Patients with Class III heart function of New York Heart Association Functional Classification (NYHA) or higher upon the Investigators evaluation.
* Patients with pulmonary dysfunction upon the Investigator's evaluation.
* Patients who have undergone Endoscopic Retrograde Cholangiopancreatography (ERCP) or have a history of cholecystitis or liver abscess.
* Patients with a duodenal ulcer, gastric ulcer, or previous and existing pancreatitis.
* Patients with gallstones (diameter ≥ 20 mm) with clinical symptoms.
* Patients with on-going thyroid dysfunction, not stabilized despite appropriate treatment.
* Patients with hemorrhage or potential hemorrhage in the digestive tract.
* Patients with gastrointestinal tract anomalies, such as gastrointestinal tract atresia, or other conditions that would result in failed placement in the gastrointestinal tract.
* Patients with a history of bowel obstruction or related diseases in the past year.
* Patients with a history of systemic lupus erythematosus or scleroderma.
* Patients with severe infections that are not controlled.
* Patients with poor general condition and having endoscopic contraindications (as evaluated by the Investigator).
* Pregnant women or planning to become pregnant.
* Patients with an alcohol dependence or substance abuse.
* Patients with unstable psychiatric disorders.
* Patients who are enrolled in another investigational study and have not completed the required follow-up period.
* Patients with an allergy to any of the components of the investigational device.
* Presence of helicobacter pylori resistant to medical treatment.
* Patients with any other conditions evaluated by the Investigators as unsuitable for participating in the clinical investigation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2025-02-02 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Performance（EFFICACY） Endpoint: | 3 months after device implantation procedure
  1) Extra weight loss percentage (EWL%) at 3 months after device implantation procedure.

SECONDARY OUTCOMES:
Use abdominal X-ray evaluate Device implantation status | V1-V5(90±7 days)
  Abdominal X-ray will be performed 1 month after the implantation procedure (Visit 4) and before Gastric Bypass Stent retrieval (Visit 5). An abdominal plain film will be used to assess the status of the Gastric Bypass Stent.
  1. The stent is completely located in the duodenal bulb.
  2. The stent is unfolded, and the outline is clear.
Performance（EFFICACY） Endpoint: | 1, 3, 4, 6, and 9 months after the procedure.
  BMI change from baseline at 1, 3, 4, 6, and 9 months after the procedure.
Performance（EFFICACY） Endpoint: | 3, 6, and 9 months after the procedure.
  Changes in glycated hemoglobin (HbA1c) at 3, 6, and 9 months after the procedure.
Performance（EFFICACY） Endpoint: | at 1, 3, 4, 6, and 9 months after the procedure.
  Drug dose of hypoglycemic agents at 1, 3, 4, 6, and 9 months after the procedure.
Changes in blood glucose-related indicators of the patients from Baseline | from baseline to 1, 3, 4, 6, and 9 months after the procedure.
  Through observe the changes of (fasting insulin, fasting blood glucose, fasting C-peptide) from baseline to 1, 3, 4, 6, and 9 months to evaluate whether implanting the investigational device will bring any changes to patients' blood glucose.
Performance（EFFICACY） Endpoint: | from baseline to 3, 4, 6, and 9 months after the procedure.
  Difference in blood lipid (total cholesterol [TC], triglyceride [TG], high density lipoprotein C [HDL-C], low-density lipoprotein C [LDL C]) change from baseline to 3, 4, 6, and 9 months after the procedure.
Satisfaction assessed by the quality of life questionnaire (BQL) | from baseline to 9 months after the procedure.
  The bariatric quality of life (BQL) questionnaire will be used to measure subject quality of life. The BQL contains 13 items rated on a scale of 1 to 5 (Absolutely wrong to Absolutely right, respectively). The maximum total score is 65, with a higher score indicating a higher quality of life. BQL total scores will be recorded in the eCRF to evaluate patients' life quality before and after percudure.
Satisfaction assessed by the visual analog scale (VAS) scale | VAS scale will be assessed before and after procedure，from baseline to 1, 3, 4, 6, and 9 months after the procedure.
  The visual analog scale (VAS) is a tool widely used to measure subject-reported pain intensity. It is a 10cm long ruler, with a "0" end and a "10" end, with 0 indicating no pain and 10 indicating the worst possible pain in subject's imagination.

OTHER OUTCOMES:
Occurrence numbers of the Clinically significant changes of laboratory tests throughout the clinical investigation. | Through out the whole study V1-V8(9 months after the procedure)
  Collect the numbers of the Clinically significant changes of laboratory tests based on investigator's evaluation to the lab tests result before and after procedure.
Occurrence numbers of complications associated with the investigational device and the procedure. | Through out the whole study V1-V8(9 months after the procedure)
  Collect the complications associated with the investigational device and the procedure based on investigator's clincial judgement.

IPD SHARING:
Plan to Share IPD: No